CLINICAL TRIAL: NCT05714774
Title: Evaluation of Different Methods of Ultrasound Image Analysis for Real-time Monitoring of HIFU Prostate Cancer Treatment Feasibility Study
Brief Title: Evaluation of Different Methods of Ultrasound Image Analysis for Real-time Monitoring of HIFU Prostate Cancer Treatment
Acronym: ELASTO-US
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL22_0522; 2022-A01958-35 (Other: IDRCB)
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; HIFU; Focal One; Prostate cancer; focal treatment; total ablation; hemi ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with localized prostate cancer (Experimental): Patients with localized prostate cancer for which focal treatment, hemi-ablation or total ablation of the prostate is indicated will be treated by HIFU applied by FocalOne device.
  Interventions: Device: HIFU treatment of prostate cancer

INTERVENTIONS:
Device: HIFU treatment of prostate cancer — HIFU treatment using Focal One (EDAP TMS) combined with the acquisition of additional ultrasound images before, between, and after HIFU shots will be performed.

SUMMARY:
The ELASTO-US study is a single center feasibility study to evaluate 3 methods of analyzing real-time ultrasound images acquired during High Intensity Focused Ultrasound (HIFU) treatment in patients with localized prostate cancer.

Real-time ultrasound acquisitions will be programmed at specific times and recorded during HIFU treatment. At the end of the treatment, these recordings will be exported in an anonymized way and analyzed according to the 3 different methods.

A multiparametric-MRI will be performed in addition to the usual practice within 5 days after the treatment in order to control the area necroticised by the treatment. The mp-MRI will be the reference method against which the results obtained by the 3 methods of ultrasound image analysis will be compared.

Techniques capable of providing safe and robust information on the progress of HIFU-generated necrosis would greatly limit the risks of overtreatment that can lead to side effects such as urinary incontinence as well as the risks of under treatment that can lead to cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has been clearly informed of the study and has agreed, with sufficient time for reflection, to participate by signing the study informed consent form.
* Male aged ≥ 50 years,
* PSA ≤ 15 ng/mL
* diagnosis of localized prostate cancer (stage T1 or T2) with a Gleason score of ≤ 7
* Focal, hemiablation or ablation HIFU treatment validated in Multidisciplinary Concerted Meeting
* Patient enrolled in Medicare or equivalent plan.
* Interpretable preoperative multiparametric MRI performed within 180 days prior to surgery

Exclusion Criteria:

* an ASA score >3
* brachytherapy for prostate cancer
* Person of full age protected by law (person under guardianship or curatorship).
* Contraindication to HIFU treatment as defined in the Focal One instructions for use : - Multiple intraprostatic calcifications inducing, on ultrasound, a shadow cone in the prostate preventing the penetration of ultrasound and therefore the realization of the treatment.
* Presence of permanent radioactive implants in the rectal wall.
* Presence of an implant (stent, catheter) located less than 1 cm from the treatment area.
* Fistula of the urinary tract or rectum.
* Anal or rectal fibrosis, anal or rectal stenosis or other abnormalities making insertion of the Focal One® catheter difficult.
* Anatomical abnormality of the rectum or rectal mucosa.
* Patient with an artificial sphincter, penile prosthesis or intraprostatic implant, such as a stent.
* History of inflammatory bowel disease.
* Current urogenital infection (infection should be treated prior to HIFU treatment).
* Patient allergic to latex with known severe reactionsCounter-indications to anesthesia

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
The percentage of analyses that could be completed for each of the three HIFU necrosis detection techniques | At day 0
  To determine the feasibility of implementing the Gray Level Histogram, The Nakagami imaging and proposed in this study, different factors will take into account : the quality of the acquired ultrasound images, the quality of the ultrasound image registration and the quality of the MRI image registration.
  The implementation of passive elastography, one of the three new methods proposed in this study, requires the presence of a sufficient wavefield in the tissue under study. An ultrasound expert will evaluate this aspect and determine whether or not the mechanical properties of the tissue can be assessed by passive elastography.

SECONDARY OUTCOMES:
To determinate the threshold to differenciate the necrotic area from the non necrotic area | at the latest on day 5 after HIFU treatment
  The threshold of the necrotic area will be determined by optimizing the sensitivity/specificity between voxels (necrotic, partially necrotic or non-necrotic).
  On post-op MRI, the prostate volume will be cut into voxels where each voxel will be classified according to its level of necrosis (total, partial or non-necrotic) by an expert radiologist.
To determinate the threshold to differenciate the partially necrotic area from the non necrotic area | at the latest on day 5 after HIFU treatment
  The threshold of the necrotic area will be determined by optimizing the sensitivity/specificity between voxels (necrotic, partially necrotic or non-necrotic).
  On post-op MRI, the prostate volume will be cut into voxels where each voxel will be classified according to its level of necrosis (total, partial or non-necrotic) by an expert radiologist.
To compare the segmentation of the necrotic zone obtained with the studied parameter to the segmentation obtained with the post treatment MRI | at the latest on day 5 after HIFU treatment
  The Hausdorff distance, which evaluates the similarity with necrotic areas on post-op MRI, will be calculated for each parameter, for each patient and for each of the two segmentation modalities. A total of 12 Hausdorff distances per patient.
To compare the segmentation of the partially necrotic zone obtained with the studied parameter to the segmentation obtained with the post treatment MRI. | at the latest on day 5 after HIFU treatment
  The Hausdorff distance, which evaluates the similarity with necrotic areas on post-op MRI, will be calculated for each parameter, for each patient and for each of the two segmentation modalities. A total of 12 Hausdorff distances per patient.
To assess of the impact of patient characteristics and treatment history for prostate cancer. | at the latest on day 5 after HIFU treatment
  The segmentations obtained with the studied parameter will be analyzed with respect to the following patient characteristics:
  * Pre-treatment prostate volume.
  * Treatment strategy (focal, hemi or total ablation)
  * Treatment history (primary or retreatment)
  * Possible associated surgical procedures (TURP, incision, ...)
  * Gleason score of the tumor
To assess of the tolerance | at the latest on day 5 after HIFU treatment
  The tolerance of the treatment will be evaluated by recording the adverse events that occurred during the patient follow-up with regard to the prolongation of the anaesthesia (approximately 20 minutes) and the realization of the mp MRI with postoperative contrast injection

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Crouzet, Pr, Principal Investigator — Service d'Urologie et Chirurgie de la Transplantation - Hôpital Edouard Herriot - Hospices Civils de Lyon
Locations (1):
- Service d'Urologie et Chirurgie de la Transplantation - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon, France